CLINICAL TRIAL: NCT02110303
Title: Dual Antiplatelet Therapy to Inhibit Coronary Atherosclerosis and Myocardial Injury in Patients With Necrotic High-Risk Coronary Plaque Disease
Brief Title: DIAMOND - Dual Antiplatelet Therapy to Reduce Myocardial Injury
Acronym: DIAMOND
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIAMOND-14/SS/0089
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 18F-F Positive - Ticagrelor (Experimental): Ticagrelor oral tablets, one (90mg) tablet, twice daily, 12 month duration
  Interventions: Drug: Ticagrelor
- 18F-F Positive - Placebo (Placebo Comparator): Identical placebo, one tablet, twice daily, 12 month duration
  Interventions: Drug: Placebo
- 18F-F Negative - Ticagrelor (Experimental): Ticagrelor oral tablets, one (90mg) tablet, twice daily, 12 month duration
  Interventions: Drug: Ticagrelor
- 18F-F Negative - Placebo (Placebo Comparator): Identical placebo, one tablet, twice daily, 12 month duration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor — oral, 90mg tablets, twice daily, 12 month duration
  Other Names: Brilique; Brilinta; Possia; AZD6140; SUB30898; B01AC24
  Arms: 18F-F Negative - Ticagrelor; 18F-F Positive - Ticagrelor
Drug: Placebo — Oral tablet (identical to ticagrelor), twice daily, 12 month duration
  Arms: 18F-F Negative - Placebo; 18F-F Positive - Placebo

SUMMARY:
Heart attacks are most commonly caused by rupture of fatty deposits (plaques) within the wall of heart blood vessels. It appears that this process can also frequently occur without causing any symptoms and these events likely explain the development of narrowing within the heart arteries which can subsequently produce symptoms of angina (chest pain).

Previous research has shown a specialised scanner known as a PET (positron emission tomography) scan can identify these recently ruptured plaques in patients without symptoms of a heart attack and these patients have changes on a blood test (troponin) which suggest that they are at higher risk of having a heart attack in the future. This study aims to identify these patients using the PET scan and then see if the markers of increased heart attack risk can be reduced by the use of a blood thinning medication (ticagrelor) which is already a well recognised treatment for people who have suffered a recent heart attack.

DETAILED DESCRIPTION:
The investigators aim to recruit patients with multivessel, clinically stable coronary artery disease. Patients will undergo baseline investigations including CT-PET imaging using 18F-Sodium Fluoride (18F-F) tracer to detect potentially unstable coronary plaques. The groups will be separated into those with and without 18F-F uptake. Each of these groups will be randomised to receive oral ticagrelor or a matched placebo in addition to their usual medications. Patients will remain on aspirin but will not be eligible for the trial if taking additional antiplatelet/anticoagulant treatments. The treatment will be continued for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years with angiographically proven multivessel coronary artery disease defined as at least two major epicardial vessels with any combination of either (a) >50% luminal stenosis, or (b) previous revascularization (percutaneous coronary intervention or coronary artery bypass graft surgery).
* Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

* An acute coronary syndrome within the last 12 months
* An indication for dual anti-platelet therapy, such as drug eluting stent
* Inability to take aspirin
* Receiving thienopyridine therapy such as clopidogrel or prasugrel
* Percutaneous coronary intervention or coronary artery bypass graft surgery within the last 3 months
* Inability or unwilling to give informed consent
* Woman with child-bearing potential and who are breastfeeding will not be enrolled into the trial (woman who have experienced menarche, are pre-menopausal, have not been sterilised or who are currently pregnant)
* Known hypersensitivity to ticagrelor or one of its excipients
* Active pathological bleeding or bleeding diathesis
* Significant thrombocytopenia: <100 x 10^9 /L
* History of intracranial haemorrhage
* Moderate to severe liver impairment (Child's Grade B or C)
* Maintenance therapy with strong cytochrome P450 3A4 (CYP3A4) inhibitors, such as ketoconazole, nefazodone, ritonavir, indinavir, atazanavir, or clarithromycin
* Major intercurrent illness or life expectancy <1 year
* Renal dysfunction (eGFR ≤30 mL/min/1.73 m2)
* Contraindication to iodinated contrast agents
* Planned coronary revascularization or major non-cardiac surgery in the next 12 months
* Maintenance therapy with simvastatin at doses greater than 40mg daily
* Receiving oral anticoagulants including warfarin, rivaroxaban, dabigatran or apixaban.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05-26 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Plasma high sensitivity cardiac troponin I (hsTnI) concentration in patients with coronary 18F-fluoride uptake. | 30 days

SECONDARY OUTCOMES:
Plasma hsTnI concentrations in patients without coronary 18F-fluoride uptake. | 30 days
High sensitivity cardiac troponin I (hsTnI) concentration in total study population. | 30 days
Plasma high-sensitivity troponin (hsTnI) concentration | 1 year
  In total population and in 18F-F PET positive and negative sub-groups
Calcium score and plaque volume at the site of baseline coronary 18F-fluoride uptake | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David E. Newby, PhD, Study Chair — University of Edinburgh; Philip D. Adamson, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Edinburgh Heart Centre, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999
- [Background] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Derived] Doris MK, Meah MN, Moss AJ, Andrews JPM, Bing R, Gillen R, Weir N, Syed M, Daghem M, Shah A, Williams MC, van Beek EJR, Forsyth L, Dey D, Slomka PJ, Dweck MR, Newby DE, Adamson PD. Coronary 18F-Fluoride Uptake and Progression of Coronary Artery Calcification. Circ Cardiovasc Imaging. 2020 Dec;13(12):e011438. doi: 10.1161/CIRCIMAGING.120.011438. Epub 2020 Dec 10. PMID 33297761
- [Derived] Moss AJ, Dweck MR, Doris MK, Andrews JPM, Bing R, Forsythe RO, Cartlidge TR, Pawade TA, Daghem M, Raftis JB, Williams MC, van Beek EJR, Forsyth L, Lewis SC, Lee RJ, Shah ASV, Mills NL, Newby DE, Adamson PD. Ticagrelor to Reduce Myocardial Injury in Patients With High-Risk Coronary Artery Plaque. JACC Cardiovasc Imaging. 2020 Jul;13(7):1549-1560. doi: 10.1016/j.jcmg.2019.05.023. Epub 2019 Aug 14. PMID 31422134
- [Derived] Moss AJ, Doris MK, Andrews JPM, Bing R, Daghem M, van Beek EJR, Forsyth L, Shah ASV, Williams MC, Sellers S, Leipsic J, Dweck MR, Parker RA, Newby DE, Adamson PD. Molecular Coronary Plaque Imaging Using 18F-Fluoride. Circ Cardiovasc Imaging. 2019 Aug;12(8):e008574. doi: 10.1161/CIRCIMAGING.118.008574. Epub 2019 Aug 6. PMID 31382765

DOCUMENTS (2):
  • Study Protocol (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT02110303/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT02110303/SAP_001.pdf